CLINICAL TRIAL: NCT00378833
Title: A Worldwide, Multicenter, Double-Blind, Parallel Study to Evaluate the Tolerability of MK0524A Versus Niacin Extended-Release
Brief Title: Tolerability of MK0524A Versus Niacin Extended-Release (0524A-054)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524A-054; 2006_529
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Hypercholesterolemia; Hyperlipidemia
Keywords: Primary Hypercholesterolemia or Mixed Hyperlipidemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Hyperlipoproteinemia Type II | interventions — Niacin; MK-0524

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: niacin (+) laropiprant — Duration of Treatment: 18 Weeks
  Other Names: MK0524A
Drug: niacin — Duration of Treatment: 18 Weeks

SUMMARY:
This is a 16-week clinical trial in lipid clinic patients for whom niacin therapy is appropriate to evaluate the tolerability of MK0524A versus niacin extended-release. There will be 6 scheduled clinic visits and 2 treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient is an appropriate candidate for niacin therapy (at risk for heart disease) and triglycerides < 500 mg/dL

Exclusion Criteria:

* Patients with a history of any cardiovascular event directly linked to atherosclerosis with a low density lipoprotein-cholesterol (LDL-C) >/= 130 mg/dL and/or not on a statin
* Patients with diabetes and LDL-C >/= 130 mg/dL. Patients with >/= 2 heart disease risk factors and LDL-C >/= 160 mg/dL.
* Patients who have had a cardiovascular event (e.g., heart attack, stroke) within the previous 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Actual)
Dates: Start 2006-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Global Flushing Severity Score (GFSS) over 16 weeks

SECONDARY OUTCOMES:
Safety/tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Maccubbin D, Koren MJ, Davidson M, Gavish D, Pasternak RC, Macdonell G, Mallick M, Sisk CM, Paolini JF, Mitchel Y. Flushing profile of extended-release niacin/laropiprant versus gradually titrated niacin extended-release in patients with dyslipidemia with and without ischemic cardiovascular disease. Am J Cardiol. 2009 Jul 1;104(1):74-81. doi: 10.1016/j.amjcard.2009.02.047. PMID 19576324
- Available data/document: CSR synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html